CLINICAL TRIAL: NCT04403776
Title: A Phase 1, Randomized, Open-Label, 2-Way Crossover Study To Evaluate Single Dose And Steady State PK And Bioavailability Between A Modified Release Tofacitinib (11 Mg QD) And The Immediate Release Tofacitinib (5 Mg BID) In Chinese Healthy Subjects
Brief Title: PK and Bioavailability Comparison of Tofacitinib Between a Modified Release and The Immediate Release Formulation
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A3921213
Record Dates: First submitted 2020-05-04; First posted 2020-05-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of the two treatment sequences. Each treatment sequence will consist of two periods, separated by a washout phase of no less than 72 hours from the AM dose on Day 7.
  Treatment A (Test): Single oral dose of tofacitinib MR 11 mg, administered as 1 x MR 11 mg tablet, in a fasting state on Day 1 followed by once daily dosing (QD) on Days 3, 4, 5, 6 and 7.
  Treatment B (Reference): Two separate oral doses (12 hours apart) of tofacitinib IR 5 mg, administered one in the morning in a fasting state and one in the evening at least 2 hours after dinner on Day 1 followed by 5 mg IR every 12 hours on Days 3, 4, 5, 6 and 7.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Treatment A, separated washout phase, followed Treatment B. (Experimental): Treatment A:
  Single oral dose of tofacitinib MR 11mg, administered as 1xMR 11mg tablet, in a fasting state on Day 1 followed by once daily dosing (QD) on Days 3, 4, 5, 6 and 7.
  washout phase: no later than 72 hours
  Treatment B:
  Two separate oral doses (12 hours apart) of tofacitinib IR 5mg, administered one in the morning in a fasting state and one in the evening at least 2 hours after dinner on Day 1 followed by 5 mg IR every 12 hours on Days 3, 4, 5, 6 and 7.
  Interventions: Drug: tofacitinib MR 11 mg; Drug: tofacitinib IR 5 mg
- Treatment B, separated washout phase, followed Treatment A. (Experimental): Treatment A:
  Single oral dose of tofacitinib MR 11mg, administered as 1xMR 11mg tablet, in a fasting state on Day 1 followed by once daily dosing (QD) on Days 3, 4, 5, 6 and 7.
  Washout phase: no later than 72 hours
  Treatment B:
  Two separate oral doses (12 hours apart) of tofacitinib IR 5mg, administered one in the morning in a fasting state and one in the evening at least 2 hours after dinner on Day 1 followed by 5 mg IR every 12 hours on Days 3, 4, 5, 6 and 7.
  Interventions: Drug: tofacitinib MR 11 mg; Drug: tofacitinib IR 5 mg

INTERVENTIONS:
Drug: tofacitinib MR 11 mg — Single oral dose of tofacitinib MR 11 mg, administered as 1 x MR 11 mg tablet, in a fasting state on Day 1 followed by once daily dosing (QD) on Days 3, 4, 5, 6 and 7.
Drug: tofacitinib IR 5 mg — Two separate oral doses (12 hours apart) of tofacitinib IR 5 mg, administered one in the morning in a fasting state and one in the evening at least 2 hours after dinner on Day 1 followed by 5 mg IR every 12 hours on Days 3, 4, 5, 6 and 7.

SUMMARY:
A study to characterize the single-dose and steady-state pharmacokinetics of tofacitinib Modified Release (MR) formulation as well as to compare the extent of absorption of the MR 11 mg formulation (once daily) to that of the Immediate Release (IR) 5 mg formulation (twice daily) of tofacitinib in Chinese healthy subjects under fasted conditions.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be of Chinese ethnicity (individuals currently residing in mainland China who were born in China and have both parents of Chinese descent).
* Healthy male and/or female subjects of non-childbearing potential
* Female subjects of non-childbearing potential must meet at least one of the following criteria:
* Achieved postmenopausal status, defined as follows: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level confirming the postmenopausal state;
* Have undergone a documented hysterectomy and/or bilateral oophorectomy;
* Have medically confirmed ovarian failure.
* Body Mass Index (BMI) of 19.0 to 26.0 kg/m2; and a total body weight >50 kg (110 lbs).

Exclusion Criteria:

Subjects presenting with any of the following will not be included in the study:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Clinically significant infections within the past 3 months prior to first dosing (eg, those requiring hospitalization or parenteral antibiotics, or as judged by the Investigator), evidence of any infection within the past 7 days prior to first dosing, history of disseminated herpes simplex infection or recurrent (>1 episode) or disseminated herpes zoster.
* Any condition possibly affecting drug absorption (eg, gastrectomy, colon resection, etc.).
* Use of CYP3A4 inhibitors (eg, ketoconazole, ciprofloxacin, diltiazem) or inducers (eg, phenytoin, carbamazepine, rifampin) within 14 days or 5 half lives (whichever is longer) prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2019-02-12 (Actual); Study Completion 2019-02-12 (Actual)

PRIMARY OUTCOMES:
Area under the plasma concentration time profile from time zero extrapolated to infinite time (AUCinf) | Plasma PK samples will be collected pre dose and after the Day 1 AM dose of MR and IR treatments and the PM dose of the IR treatment.
Area under the plasma concentration time profile from time zero to the time of the last quantifiable concentration (AUClast) | Plasma PK samples will be collected pre dose and after the Day 1 AM dose of MR and IR treatments and the PM dose of the IR treatment.
Area under the concentration time profile for the 24 hour period (AUC24) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)

SECONDARY OUTCOMES:
Single-dose PK: maximum observed concentration (Cmax) | Plasma PK samples will be collected pre dose and after the Day 1 AM dose of MR and IR treatments and the PM dose of the IR treatment.
Single-dose PK: time for Cmax (Tmax) | Plasma PK samples will be collected pre dose and after the Day 1 AM dose of MR and IR treatments and the PM dose of the IR treatment.
Single-dose PK: terminal half-life (t1/2) | Plasma PK samples will be collected pre dose and after the Day 1 AM dose of MR and IR treatments and the PM dose of the IR treatment.
Single-dose PK: area under the plasma concentration-time profile from time 0 to tau (AUCtau) | Plasma PK samples will be collected pre dose and after the Day 1 AM dose of MR and IR treatments and the PM dose of the IR treatment.
Steady-state PK: Cmax | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: lowest concentration observed (Cmin) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: average concentration (Cav) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: Tmax | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: concentration at 24 hours (C24) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: peak to trough ratio (PTR) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: peak to trough fluctuation (PTF) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: peak to trough swing (PTS) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: observed accumulation ratio for AUC (Rac) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Steady-state PK: observed accumulation ratio for Cmax (Rac,Cmax) | Blood samples for assessing steady state PK will be collected prior to dosing on Days 5, 6 and 7 and after dosing on Day 7 (up to 24 hours post Day 7 AM dose)
Number (%) of subjects with treatment-emergent adverse events | approximately 18 days
  ECG, Clinical Laboratories, Vitals Signs and Physical Exams will be used as a safety measure to detect any AEs.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Shuguang Hospital Affiliated to Shanghai University of TCM/Phase I Unit, Shanghai, China

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=A3921213